CLINICAL TRIAL: NCT06487221
Title: A Phase II Trial of Avutometinib in Combination With Defactinib in Metastatic Diffuse Gastric Cancer
Brief Title: Avutometinib and Defactinib in Diffuse Gastric Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ryan H. Moy, MD, PhD (Other)
Collaborators: Verastem, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Ryan H. Moy, MD, PhD, Assistant Professor of Medicine, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAV0009
Record Dates: First submitted 2024-06-26; First posted 2024-07-05 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Gastric Cancer; Stomach Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — defactinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Avutometinib & Defactinib (Experimental): Avutometinib: Study participants will receive Avutometinib 3.2mg orally two times per week for three weeks in a row followed by one week of rest
  Defactinib: Study participants will receive Defactinib 200mg twice daily for three weeks in a row followed by one week of rest
  Interventions: Drug: Avutometinib; Drug: Defactinib

INTERVENTIONS:
Drug: Avutometinib — 3.2mg orally
  Other Names: VS6766
Drug: Defactinib — 200 mg orally
  Other Names: VS-6063

SUMMARY:
The purpose of this study is to determine if the combination study treatment with avutometinib and defactinib will prolong life in participants, is effective in decreasing the size of the tumor(s), and if it is safe in subjects with diffuse-type stomach cancer.

DETAILED DESCRIPTION:
There are two main types of stomach cancer based on the appearance under the microscope: intestinal-type and diffuse-type. Some stomach cancers also have a mix of intestinal-type and diffuse-type (mixed type). The participants are being invited to take part in this research study due to having been diagnosed with stomach cancer that has spread to other parts of the body and/or cannot be surgically removed, has diffuse-type or mixed type cells or has gene changes that are associated with diffuse-type stomach cancers (such as mutations in the genes called CDH1 or RHOA), and have already been treated with chemotherapy and the disease is now growing. Defactinib is an oral drug that inhibits the protein focal adhesion kinase (FAK), which has been shown to promote growth of gastric cancer. Avutometinib (also known as VS-6766) is an oral drug that blocks an important signaling pathway in cancer cells known as the MAP kinase pathway. Avutometinib inhibits two proteins in the MAPK kinase pathway, RAF and MEK. The purpose of this study is to determine if the combination study treatment with defactinib and avutometinib is effective in improving the length of time after the start of treatment in which a participant is alive and their cancer does not grow or spread.

ELIGIBILITY:
Inclusion Criteria:

1. Histologic or cytologic evidence of gastric/gastroesophageal junction carcinoma, classified as diffuse type, poorly cohesive, signet ring cell, or mixed type. Patients with known pathogenic CDH1 and/or RHOA mutations will be allowed regardless of histology.
2. Prior therapy with at least one line of therapy for unresectable/metastatic disease, which must include platinum and fluoropyrimidine.
3. ECOG performance status of 0 or 1
4. Age ≥ 18 years
5. Adequate organ function, defined by the following laboratory parameters:

   a. Adequate hematologic function, including hemoglobin [Hb] ≥ 9.0 g/dL; platelets ≥ 100,000/mm3; and absolute neutrophil count [ANC] ≥ 1500/mm3. If a red blood cell transfusion or erythropoiesis-stimulating agent has been administered the Hb must remain stable and ≥ 9 g/dL for at least 1 week prior to first dose of study intervention.

   (i) Subjects with Hgb ≥ 8.5 g/dL and <9.0 g/dL are eligible if there is no history of significant cardiovascular risk features as per the investigator (i.e., prior myocardial infarction) b. Adequate hepatic function: (i) total bilirubin ≤ 1.5 × upper limit of normal [ULN] for the institution; patients with Gilbert syndrome may enroll if total bilirubin is < 3.0 mg/dL (51 μmol/L); (ii) alanine aminotransferase (ALT) and aspartate aminotransferase (AST)

   ≤ 2.5 × ULN (or < 5 x ULN in patients with liver metastases). c. Adequate renal function with creatinine clearance rate of ≥ 50 mL/min, as calculated by the Cockcroft-Gault formula d. International normalized ratio (INR) ≤ 1.5 and partial thromboplastin time (PTT) ≤ 1.5 x ULN in the absence of anticoagulation or therapeutic levels in the presence of anticoagulation.

   e. Albumin ≥ 3.0 g/dL (451 μmol/L). f. Creatine phosphokinase (CPK) ≤ 2.5 x ULN. g. Adequate cardiac function with left ventricular ejection fraction ≥ 55% by echocardiography (ECHO) or multiple-gated acquisition (MUGA) scan.
6. Disease that can be evaluated radiographically, which can be measurable disease or non-measurable disease per RECIST 1.1. All radiology studies must be performed within 28 days prior to start of study-directed therapy.
7. Tumor that is amenable to fresh biopsy, which may include malignant ascites that is amenable for paracentesis.
8. Baseline QTc interval < 460 ms for females and ≤ 450 ms for males (average of triplicate readings) using Fredericia's QT correction formula. NOTE: This criterion does not apply to subjects with a right or left bundle branch block.
9. Adequate recovery from toxicities related to prior treatments to at least Grade 1 by CTCAE v 5.0. Exceptions include alopecia and peripheral neuropathy grade ≤ 2. Subjects with other toxicities that are stable on supportive therapy may be allowed to participate with prior approval from the principal investigator.
10. The effects of the study drugs on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (see Section 7.6 for Contraception Guidance) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 3 months after the last dose of the study drug.
11. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Systemic anti-cancer therapy within 3 weeks of the first dose of study therapy, or within 5 half-lives of the previous drug, whichever is shorter.
2. Patients currently receiving any other investigational agent.
3. Subjects may not have had a history of malignancy other that esophagogastric cancer within two years prior to screening, with the exception of those with a negligible risk of metastasis or death (e.g., 5-year overall survival >90%) such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or stage I uterine cancer.
4. Major surgery within 4 weeks or palliative radiotherapy within 1 week of the first dose of study therapy.
5. Treatment with warfarin. Subjects on warfarin for DVT/PE can be converted to low- molecular-weight heparin (LMWH).
6. History of treatment with a direct and specific inhibitor of FAK, MEK, or KRAS.
7. Patients who had exposure to medications (with or without prescriptions), supplements, herbal remedies, or foods with potential for drug-drug interactions with avutometinib and/or defactinib within 14 days prior to the first dose of study intervention and during the course of therapy, including:

   1. Strong CYP3A4 inhibitors or inducers.
   2. Strong CYP2C9 inhibitors or inducers.
   3. Strong P-glycoprotein (P-gp) inhibitors or inducers
   4. Strong breast cancer resistance protein (BCRP) inhibitors or inducers
8. Symptomatic brain metastases requiring steroids or other local interventions. Subjects with previously diagnosed brain metastases are eligible if they have completed their treatment and have recovered from the acute effects of radiation therapy or surgery prior to study entry, have discontinued corticosteroid treatment for these metastases for at least 4 weeks prior to first dose of study therapy, and are neurologically stable.
9. Known hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) infection that is active and/or requires therapy. HIV patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with the investigational agents.
10. Active skin disorder that has required systemic therapy within the past 1 year.
11. History of rhabdomyolysis.
12. Concurrent ocular disorders including the following:

    1. Patients with history of glaucoma, history of retinal vein occlusion (RVO), predisposing factors for RVO, including uncontrolled hypertension, uncontrolled diabetes.
    2. Patients with history of retinal pathology or evidence of visible retinal pathology that is considered a risk factor for RVO, intraocular pressure > 21 mm Hg as measured by tonometry, or other significant ocular pathology, such as anatomical abnormalities that increase the risk for RVO.
    3. Patients with active or chronic, visually significant corneal disorders, other active ocular conditions requiring ongoing therapy or clinically significant corneal disease that prevents adequate monitoring of drug-induced keratopathy. Examples of visually significant corneal disorders include corneal degeneration, active or recurrent keratitis, and other forms of serious ocular surface inflammatory conditions. Visually significant corneal disorders do NOT include dry eyes, blepharitis, and uncomplicated corneal erosions.
13. Concurrent congestive heart failure, prior history of class III/IV cardiac disease (New York Heart Association [NYHA]), myocardial infarction within the last 6 months, unstable arrhythmias, unstable angina or severe obstructive pulmonary disease.
14. Inability to swallow oral medications.
15. History of hypersensitivity to any of the inactive ingredients (hydroxylpropylmethylcellulose, mannitol, magnesium stearate) of the investigational product.
16. Female subjects who are pregnant or breastfeeding. Pregnant women are excluded from this study because the risk for teratogenic or abortifacient effects with the investigational agents is unknown. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother, breastfeeding should be discontinued if the mother is treated with the investigational agents.
17. Any other medical condition (e.g., cardiac, gastrointestinal, pulmonary, psychiatric, neurological, genetic, etc.) that in the opinion of the investigator would place the subject at unacceptably high risk for toxicity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2024-10-28 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2029-05-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) Rate | 6 months
  To determine the efficacy of combination defactinib and avutometinib in patients with metastatic diffuse gastric cancer (DGC) as measured by 6-month progression-free survival (PFS) rate. PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | 6 months
  Overall response rate (ORR) defined as partial response (PR) + complete response (CR) according to Response Evaluation Criteria in Solid Tumors version 1.1 [RECIST 1.1]. PR is at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. CR is a disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
Median Progression-Free Survival | 24 months
  To determine the impact of combination defactinib and avutometinib on other measures of efficacy off progression free survival (PFS). Time from the start of treatment until disease progression or death, whichever comes first.
Median Overall Survival (OS) | Up to 5 years
  Overall survival defined as the time from the start of treatment until death or last follow-up.
Disease Control Rate (DCR) | 24 months
  DCR defined as Complete Response (CR)+ Progressive Disease (PD)+ Stable Disease (SD) as assessed per RECISIT 1. CR is a disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PD is at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions). SD is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Duration of response (DOR) | 24 months
  The duration of overall response is measured from the time measurement criteria are met for CR (Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm) or PR (At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters), whichever is first recorded, until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started).

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Moy, MD, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States